CLINICAL TRIAL: NCT00498979
Title: Phase I Evaluation of Sodium Stibogluconate in Combination With Interferon α-2b Followed by Cisplatin, Vinblastine and Dacarbazine for Patients With Melanoma or Malignancies Potentially Responsive to SSG and/or Interferons
Brief Title: Sodium Stibogluconate and IFNa-2b Followed By CDDP, VLB and DTIC Treating Pts.With Advanced Melanoma or Other Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3Y06
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Stage IV Melanoma
Keywords: stage IV melanoma; adult anaplastic astrocytoma; adult diffuse astrocytoma; adult glioblastoma; adult giant cell glioblastoma; adult pilocytic astrocytoma; adult brain stem glioma; adult anaplastic ependymoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma; adult anaplastic oligodendroglioma; adult oligodendroglioma; mixed gliomas; recurrent adult brain tumor; recurrent melanoma; adult gliosarcoma; adult subependymal giant cell astrocytoma; adult pineal gland astrocytoma
MeSH Terms: conditions — Melanoma; Astrocytoma; Glioblastoma; Ependymoma; Glioma, Subependymal; Oligodendroglioma; Glioma; Brain Neoplasms; Gliosarcoma | interventions — Introns; Cisplatin; Antimony Sodium Gluconate; Dacarbazine; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- recombinant interferon alfa-2b (Experimental): recombinant interferon alfa-2b
  Interventions: Biological: recombinant interferon alfa-2b; Drug: cisplatin; Drug: sodium stibogluconate; Drug: dacarbazine; Drug: vinblastine

INTERVENTIONS:
Biological: recombinant interferon alfa-2b — recombinant interferon alfa-2b
  Other Names: IFN 2b
Drug: cisplatin — recombinant interferon alfa-2b
  Other Names: CDDP
Drug: sodium stibogluconate — sodium stibogluconate
Drug: dacarbazine — dacarbazine
  Other Names: DTIC
Drug: vinblastine — vinblastine
  Other Names: VBL

SUMMARY:
RATIONALE: Sodium stibogluconate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Interferon alfa-2b may interfere with the growth of tumor cells and slow the growth of melanoma and other cancers. Drugs used in chemotherapy, such as cisplatin, vinblastine, and dacarbazine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sodium stibogluconate and interferon alfa-2b together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of sodium stibogluconate when given together with interferon alfa-2b, cisplatin, vinblastine, and dacarbazine in treating patients with advanced melanoma or other cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety of the combination of sodium stibogluconate and interferon alfa-2b with chemotherapy.
* To confirm the activity of sodium stibogluconate in augmenting cytokine effects.

Secondary

* To quantify the effects of sodium stibogluconate on interferon alfa-2b induced gene modulation and signal transduction pathways by measuring the serum soluble gene products.
* To define the effectiveness of sodium stibogluconate in inhibiting the protein tyrosine phosphatases SHP-1 and SHP-2 assayed from peripheral blood leukocytes of patients receiving sodium stibogluconate in combination with interferon alfa-2b.
* To define the pharmacokinetics of sodium stibogluconate in serum at escalating doses.
* To assess clinical response to the combination of sodium stibogluconate and interferon alfa-2b as priming for combination chemotherapy.

OUTLINE:

* Course 1: Patients receive sodium stibogluconate IV over 15 minutes on day 1 and days 15-18; interferon alfa-2b subcutaneously (SC) on days 8-12 and 15-18; cisplatin IV over 30-60 minutes and vinblastine IV on days 19 and 20; and dacarbazine. After a 2-week rest period, patients proceed to course 2.
* Course 2 and all subsequent courses: Patients receive sodium stibogluconate IV over 15 minutes and interferon alfa-2b SC on days 1-4; cisplatin IV over 30-60 minutes and vinblastine IV on days 5 and 6; dacarbazine. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.* NOTE: *Patients with stage IV disease who have no evidence of disease [NED} receive only 4 courses of therapy.

Cohorts of 6 patients receive escalating doses of sodium stibogluconate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which dose-limiting toxicity occurs (i.e., no more than 1 patient at a given dose experiences DLT).

Patients undergo blood sample collection periodically for immunological and pharmacokinetic studies. Samples are analyzed for serum soluble gene products and protein tyrosine phosphatase inhibition.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma or other malignancies

  * Must be refractory or resistant to established treatments OR have metastatic disease for which no effective therapy has been established
  * Gliomas or controlled CNS metastasis allowed

    * A CT scan or MRI must confirm stable brain metastases within 28 days of study entry
    * Patients with primary CNS malignancies refractory to other therapies are eligible
* Malignancy potentially responsive to sodium stibogluconate and/or interferon alfa-2b and combination chemotherapy
* Patients must have measurable or evaluable disease

  * Evaluable disease can include clinically or radiographically nonmeasurable tumor, specific tumor markers, or stage IV patients with no evidence of disease (NED)

PATIENT CHARACTERISTICS:

* Inclusion criteria:

  * ECOG performance status 0-2
  * Granulocytes > 1,500/μl
  * Platelets > 100,000/μl
  * Creatinine < 1.5 x upper limit of normal (ULN)
  * Bilirubin < 1.5 x ULN
  * AST and ALT < 1.5 x ULN (unless due to hepatic metastases)
  * Potassium ≤ 5.0 mmol/L
  * Magnesium ≤ 2.4 mg/dL
  * Creatinine clearance ≥ 60 cc/min
  * Ejection fraction ≥ 50%
* Exclusion criteria:

  * Pregnant or lactating women and fertile women or men unless surgically sterile or using effective contraception

    * All female patients of childbearing potential or less than 1 year postmenopausal must have a negative β-HCG pregnancy test at baseline and practice a medically acceptable method of birth control (i.e., oral contraceptives for at least 3 months, implantation of an intrauterine device for at least 2 months, or barrier methods [e.g., vaginal diaphragm, vaginal sponge, or condom with spermicidal jelly]) during and for 3 months after study initiation
  * History of atrial fibrillation, flutter, or other serious arrhythmia (excluding asymptomatic atrial or ventricular premature complexes) in the past 24 months
  * History of congestive heart failure currently requiring treatment; angina pectoris; or other severe cardiovascular disease (i.e., New York Heart Association class III or IV heart disease)
  * Baseline ECG abnormalities suggestive of cardiac conduction delay (i.e., first degree or greater atrio-ventricular block and/or complete or incomplete [QRS > 120 ms] bundle branch block)
  * Baseline ECG abnormalities suggestive of repolarization abnormalities (i.e., QTc ≥ 0.48 sec)
  * Culture positive acute infections requiring antibiotics within the past 14 days

    * Patients on long term suppressive antibiotic therapies are eligible
  * Known to be positive for HBsAg
  * Patients judged to not be psychologically prepared to understand informed consent or comply with an investigational study

PRIOR CONCURRENT THERAPY:

* Inclusion criteria:

  * Prior interferon therapy is allowed if administered ≥ 4 months ago
  * At least 3 weeks since prior major surgery, radiation therapy, or chemotherapy
* Exclusion criteria:

  * No prior treatment with interferon, sodium stibogluconate, cisplatin, vinblastine, or dacarbazine, except if given in an adjuvant setting
  * Patients with a prior history of solid organ allografts or allogeneic bone marrow transplant
  * Patients taking the following medications will not be eligible:

    * Amiodarone (Cordarone)
    * Disopyramide (Norpace)
    * Dofetilide (Tikosyn)
    * Procainamide (Procanbid or Pronestyl)
    * Quinidine (Quinaglute)
    * Sotalol (Betapace)
    * Erythromycin
    * Azithromycin (Z-pack)
    * Clarithromycin (Biaxin)
    * Pentamidine (Pentacarinat)
    * Trimethoprim-sulfamethoxazole (Bactrim)
    * Bepridil (Vascor)
    * Phenothiazines (e.g., prochlorperazine [Compazine], promethazine [Phenergan], or chlorpromazine [Thorazine])
    * Butyrophenones (e.g., Haloperidol [Haldol])
    * Risperidone (Risperdal)
    * Any other antipsychotic medication
    * Tricyclic or tetracyclic antidepressants (e.g., imipramine [Tofranil], amitriptyline [Elavil], desipramine [Norpramin], or nortriptyline [Pamelor])
    * Monoamine oxidase inhibitors
    * High-dose methadone
    * Arsenic trioxide
    * Dolasetron (Anzemet)
    * Any herbal preparations
  * Use of daily glucocorticoids except for physiological replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-05; Primary Completion 2010-05 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety of the combination of sodium stibogluconate and interferon alfa-2b with chemotherapy | 2 years

SECONDARY OUTCOMES:
Effects of sodium stibogluconate on interferon alfa-2b induced gene modulation and signal transduction pathways by measuring the serum soluble gene product | 2 years
Effectiveness of sodium stibogluconate in inhibiting the protein tyrosine phosphatases SHP-1 and SHP-2 assayed from peripheral blood leukocytes | 2 years
Pharmacokinetics of sodium stibogluconate in serum at escalating doses | 2 years
Clinical response to the combination of sodium stibogluconate and interferon alfa-2b as priming for combination chemotherapy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ernest C. Borden, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States